CLINICAL TRIAL: NCT04198597
Title: Exploring Two CBT-based Treatments as Interventions for Emotion Dysregulation in Misophonia
Brief Title: Exploring Two Treatments for Misophonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103962
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2021-12

CONDITIONS: Misophonia
MeSH Terms: conditions — misophonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unified Protocol, 2 week baseline (Experimental): Participants in this arm will complete two weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Unified Protocol, 4 week baseline (Experimental): Participants in this arm will complete four weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Process-based treatment, 2 week baseline (Experimental): Participants in this arm will complete two weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the process-based therapy. Process-based therapy is a flexible therapy designed to teach skills that help people manage difficult experiences. Patient and therapist work together to determine which skills will be utilized.
  Interventions: Behavioral: Process-based Cognitive Behavioral Therapy
- Process-based treatment, 4 week baseline (Experimental): Participants in this arm will complete four weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the process-based therapy. Process-based therapy is a flexible therapy designed to teach skills that help people manage difficult experiences. Patient and therapist work together to determine which skills will be utilized.
  Interventions: Behavioral: Process-based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — Please see arm/group descriptions
  Arms: Unified Protocol, 2 week baseline; Unified Protocol, 4 week baseline
Behavioral: Process-based Cognitive Behavioral Therapy — Please see arm/group descriptions
  Arms: Process-based treatment, 2 week baseline; Process-based treatment, 4 week baseline

SUMMARY:
While the investigators continue to work on better understanding Misophonia, it is also important to identify treatments that can help people who are currently suffering. Further, it is important that the treatments provided are acceptable to the people who receive them. In this study, participants will complete one of two treatments the investigators believe can help manage symptoms of Misophonia: The Unified Protocol or process-based therapy. Both treatments will use evidence-based psychological principles (e.g., managing attention or behavior) in a flexible manner and will focus on developing skills to help reduce the distress and impairment associated with Misophonia. The aims of this study are (1) to explore the acceptability and feasibility of these treatments for individuals who experience Misophonia and (2) to examine whether these treatments help reduce symptoms associated with Misophonia.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Able to read English
* Meet criteria for interfering symptoms of misophonia
* Live in North Carolina

Exclusion Criteria:

* Under age 18
* Current mania
* Current psychotic disorder
* Current anorexia
* Presents with a condition that requires immediate prioritization in treatment (e.g., suicide planning or intent)
* Has received any treatment specifically for misophonia in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Number of patients that are satisfied with treatment as measured by the credibility and expectancy questionnaire (CEQ) | up to 20 weeks
  The CEQ is a 6-item measure that asks patients about their perceptions of treatment.
Number of patients who indicate treatment was acceptable to them (i.e., the treatment approach made sense and was perceived as reasonable) | up to 20 weeks
  This form has two questions that assess how satisfied patients were with treatment and how acceptable treatment was to them. The remaining three items are open ended questions that allow patients to provide narrative feedback about their experience in treatment.

SECONDARY OUTCOMES:
Change in misophonia symptoms as assessed by the Misophonia Questionnaire | assessed weekly, up to 24 weeks
  The Misophonia Questionnaire is a 17-item questionnaire that assesses the presence of misophonia symptoms, emotions and behaviors associated with misophonic reactions, and symptom severity. The first two subscales are rated on a scale of 0 (not at all true) to 4 (always true). These two parts are summed to produce a total score ranging from 0 - 68. The severity subscale is a single item that asks an individual to provide a rating of their sound sensitivity on a scale from 0 (no sound sensitivities) to 15 (very severe sound sensitivities).
Change in anxiety as measured by the Overall Anxiety Severity and Impairment Scale | assessed weekly, up to 24 weeks
  The Overall Anxiety Severity and Impairment Scale is a five item measure that assesses interference and distress related to the experience of anxiety. Items are scored from 0 to 4 and summed to produce a total score (ranging from 0 - 20), with higher scores indicating greater functional impairment.
Change in depression as measured by the Overall Depression Severity and Impairment Scale | assessed weekly, up to 24 weeks
  The Overall Depression Severity and Impairment Scale is a five item measure that assesses interference and distress in an individual's day-to-day life related to the experience of depression. Items are scored from 0 to 4 and summed to produce a total score (ranging from 0 - 20), with higher scores indicating greater functional impairment.
Change in anger as measured by the Clinical Anger Scale | assessed weekly, up to 24 weeks
  The Clinical Anger Scale is a 21-item measure that assesses the severity of anger-related symptoms (e.g., current anger, anger about the future).Items are scored from 0 to 3 and summed to produce a total score (ranging from 0 - 63), with higher scores indicating greater anger-related symptoms.
Number of patients who use the skills taught in treatment as measured by the Skill Use Questionnaire | assessed weekly, up to 24 weeks
  The Skill Use Questionnaire is a four-item measure that assesses the extent to which patients use the skills taught in therapy and find them to be helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rosenthal, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No